CLINICAL TRIAL: NCT04183998
Title: Trans-spinal Electrical Stimulation to Restore Upper Extremity Functions in Individuals With Traumatic Brain Injury (TBI) or Spinal Cord Injury (SCI).
Brief Title: Restorative Neuromodulation for Upper Extremity Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University of California, Los Angeles (Other); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr Monzurul Alam, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20190121002
Record Dates: First submitted 2019-11-17; First posted 2019-12-03 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Brain Injury; Cervical Spinal Cord Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tsES (Experimental): trans-spinal Electrical Stimulation (tsES)
  Interventions: Other: Trans-spinal Electrical Stimulation (tsES)

INTERVENTIONS:
Other: Trans-spinal Electrical Stimulation (tsES) — Stimulation will be achieved with two self-adhesive stimulation electrodes attached to the dorsal aspect of the neck overlying the cervical vertebrae and two self-adhesive rectangular return electrodes placed over the shoulders. Spinal motor evoked potentials (sMEP) induced by trans-spinal electrical stimulation (parameters, 1 Hz with a 0.1-1 ms pulse width and monophasic waveform) to determine recruitment profiles of proximal and distal motor pools with increasing stimulation intensity ranging from 10 to 200 milliampere. Stimulation parameters for the therapeutic stimulation will be ranged from 5-40 Hz and 20-100 milliampere.

SUMMARY:
The objective of this research study is to find the efficacy of trans-spinal electrical stimulation, a non-invasive neurostimulation method to modulate the functions of spinal cord neurocircuits, on improving upper-extremity functions such as reaching and grasping in individuals suffering with traumatic brain injury (TBI) or cervical spinal cord injury (SCI); and to find the physiological changes in the neuromuscular systems after this new intervention with high-resolution electrophysiology and biomedical imaging.

DETAILED DESCRIPTION:
Spinal cord is composed of specialized neural networks, capable of executing different functions. Although the command for upper-limb functions such as reaching and grasping is delivered from the brain, the cervical spinal cord circuits work as an important hub for not only executing the task, but also amplify the command and maintain the dynamics with proper feedback mechanisms with it's reflex circuitry. A simple reaching and grasping function requires spatiotemporal coordination of upper-limb joints and the neuromuscular systems, their adaptation and control in gravity. For human, these physiological activities are well choreographed by sets of neural networks. In combination with afferent sensory inputs, these network circuits work with the motor periphery to generate a series of motor acts during each task. Normally, the activity of these spinal networks are regulated supraspinally and by peripheral sensory inputs. In case of the loss of supraspinal inputs, resultant of a traumatic brain injury (TBI) or cervical spinal cord injury (SCI), upper-limb motor tasks maybe enabled by directly activating these specialized cervical cord networks via external stimuli. Recent studies have demonstrated that neuromodulation via spinal cord stimulation can effectively restore upper-limb motor function in patients with chronic neurological injuries.

Traumatic injuries to the central nervous system (CNS) such as TBI and SCI are devastating events leaving patients with impairment of motor, sensory and autonomic functions. Mainstay for the treatment is still limited to rehabilitation by physical therapy and training. In few patients, however, neuroplasticity and repair mechanisms are considered to contribute to recovery of paresis in the acute stage of the injury and stops in the chronic stage. But, three recent groundbreaking pilot studies have shown that the recovery can be further amplified in the chronic stage by the novel treatment of trans-spinal electrical stimulation. However, the rehabilitation related to this recovery is not well understood, and thus it is a challenge to be convinced with the efficacy of this new therapy. A deeper understanding of the physiology in a larger trial of two different but related neurological patient groups, proposed in this study, will significantly help the researcher to prove the efficacy and understand the mechanism of trans-spinal electrical stimulation therapy for the patients. This study will further assist the researchers to design even a better therapeutic intervention for neurological impaired patients.

ELIGIBILITY:
Inclusion Criteria:

* At least one year post-injury
* Non-progressive TBI or SCI at above C7 spinal level
* Unable to grip or reach independently, and requires assistance for daily living activities
* Spinal reflexes remain functional below the lesion
* Female participants of child-bearing potential must be on a standard method of contraception and must not be pregnant

Exclusion Criteria:

* Cardiopulmonary disease or dysfunction, high blood pressure or other medical risk factors
* Received Botox injection in the prior 6 months
* Cervical fusion with any metal which may interfere with trans-spinal electric currents
* Other electronic implants such as cardiac pacemakers, defibrillators, shunts, stents etc.
* Unhealed fracture, contracture, pressure sore, or infections
* Currently receiving treatments for either pain management or spasticity or depression

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | 12 months
  Fugl-Meyer Assessment for upper extremity will be used for the measurement of upper limb motor functional recovery. We will adobe the version of the University of Gothenburg approved by Fugl-Meyer AR. In a cumulative numerical scoring to evaluate the physical performance including coordination and speed of the upper extremities, functions of hand and wrist will be assessed separately. The test is constructed with different stages of motor recovery: 1) reflexes reoccur; 2) stereotyped volitional movement can be imitated within flexor and extensor synergies; 3) movements can be performed that deviate from primitive synergies; and 4) reflexes are normalized. A 3-point ordinal scale will be applied to each item: 0=the detail cannot be performed, 1=the detail can be partially performed; 2=the detail can be fully performed. The maximum motor score for the upper extremity can be 66 points where higher score will indicate better function.
Modified Ashworth Scale | 12 months
  Modified Ashworth Scale is a measurement tool for muscle tone which can be used to measure upper-limb spasticity at different upper extremity segments. It is a 6-point numerical scoring system: 0=no increase in muscle tone, 1=slight increase in muscle tone; 1+=slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder; 2=more marked increase in muscle tone through most of the ROM, but affected part move easily; 3=considerable increase in muscle tone, passive movement difficult; 4=affected part rigid. Lower scores after the treatment will indicate the decrease of muscle spasticity around the specific upper extremity joints, on contrary, higher scores will indicated the aggravation of the muscle spasticity of the segment.The test will be carried out before and after each of the three experimental phases (Phase 1-3).
Action Research Arm Test | 12 months
  Action Research Arm Test is also a cumulative numerical rating scale for the measurement of upper extremity performance,which is frequently used in research and clinical practice. The reliability of this test has been evaluated in several studies using reliability coefficients such as Spearman's rank correlation coefficient and intra-class correlation coefficient. This test focuses more on the hand functions with 4 basic movements: grasp, grip, pinch and gross movement, and is assessed on a 4-category ordinal scale (i.e., 0,1,2, and 3) with totally 19 items.The ordinal scale is not only related to the degree of completion of an action, but also related to the time cost:0=the motion task cannot be performed, 1=the motion task can be partially performed, 2=the motion task can be fully performed, but clunky or slow, 3=the motion task can be fully performed normally.
Wolf Motor Function Test | 12
  The Wolf Motor Function Test is a quantitative index of upper extremity motor ability examinable through the use of timed and functional tasks. The Wolf Motor Function Test has been posited as instructive for assessing the motor status of higher functioning chronic patients with stroke and traumatic brain injury, in terms of severity and upper extremity motor deficiency.It has 17 items and is assessed with two scoring systems: 1) a 5-category ordinal scale where higher scores mean better motor function; 2) time counting scale where higher scores mean slower movement and worse motor function.Grip force has also been concluded in this test.

SECONDARY OUTCOMES:
Functional Independence Measurement | 12 months
  In addition to assessing patients' post-injury functional status, the Functional Independence Measure will also be monitored once a month and in follow-up. The Functional Independence Measure is an 18-items,7-level questionnaire assessment designed to evaluate the amount of assistance required by the disabled individual to perform basic life activities safely and effectively.

OTHER OUTCOMES:
Electrophysiology | 18 months
  Muscular physiological activity will be collected via surface electromyography, mechanomyography and sonomyography of upper-limb muscles including flexor digitorum, extensor digitorum, brachioradialis, biceps brachii, and triceps brachii. Forelectromyography: Four pairs of Ag/Agl electrodes (Bluesensor, Ambu Inc. America) will be attached on to the skin surface of the muscle bellies, with a 2-cm center separation. A single reference electrode will be attached on the skin surface of olecranon. For mechanomyography and sonomyography, custom sensors form the laboratory of the Department of Biomedical Engineering, The Hong Kong Polytechnic University will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Monzurul Alam, PhD, Principal Investigator — Research Assistant Professor
Locations (1):
- Department of Biomedical Engineering, The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
On request and under condition.